CLINICAL TRIAL: NCT03582228
Title: Bridging Recovery Allies in Virtual Environments (BRAVE)-Understanding Feasibility and Acceptability of Using Virtual Environments for Social Communication in Persons With TBI
Brief Title: Bridging Recovery Allies in Virtual Environments
Acronym: BRAVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: The Institute for Rehabilitaion and Research Foundation (Other)
Responsible Party: Principal Investigator, Hilary Nicole Touchett, Doctoral Student, Robert Wood Johnson Foundation Future of Nursing Scholar, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HSC-SN-18-0491
Record Dates: First submitted 2018-06-27; First posted 2018-07-10 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Traumatic Brain Injury
Keywords: Virtual Environments; Social Communication
MeSH Terms: conditions — Brain Injuries, Traumatic; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Envrionment for Social Communication (Experimental): Once the intervention begins, participants will meet online from home for one-hour sessions twice a week (twelve sessions over six weeks).
  Weekly sessions will follow a standardized format:
  * 15 minutes- Social support group (guided discussion of experiences related to weekly topic)
  * 20 minutes- Didactic instruction
  * 15 minutes- Role playing
  * 10 minutes- Debriefing and group feedback
  Interventions: Behavioral: Virtual Envrionment for Social Communication

INTERVENTIONS:
Behavioral: Virtual Envrionment for Social Communication — Once the Virtual Envrionment for Social Communication intervention begins, participants will meet online from home for one-hour sessions twice a week (twelve sessions over six weeks).
  Weekly sessions will follow a standardized format:
  * 15 minutes- Social support group (guided discussion of experiences related to weekly topic)
  * 20 minutes- Didactic instruction
  * 15 minutes- Role playing
  * 10 minutes- Debriefing and group feedback

SUMMARY:
The Bridging Recovery Allies in Virtual Environments (BRAVE) study aims to evaluate the acceptability and feasibility of implementing a virtual environment (VE) social support group for social communication training among adults with traumatic brain injury (TBI).

ELIGIBILITY:
Inclusion Criteria:

* subjects with a traumatic brain injury
* between the age of 18 and 80
* living in the community
* able to read and speak English,
* are more than 1-year post-injury
* are accessible by phone,
* report independent computer usage over the last 6 months
* have access to a computer meeting minimum specifications for the Learning in Virtual Environments (LIVE) platform (requires Windows)
* have broadband Internet connection,
* achieve a Galveston Orientation Assessment Test (GOAT) score >75 to ensure appropriate levels of cognition for the study
* and score >93.8 on the Western Battery Aphasia-Revised (WAB-R) scale to indicate sufficient communicative abilities to participate in a social support group and exit interview group.
* able to understand and independently consent for the study and provide written consent prior to enrollment in the study

Exclusion Criteria:

- verbal communication impairments will be excluded as measured by the WAB-R, as this study intends to focus on persons with social communication deficits rather than verbal deficits.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Perceived Usability as Assessed by the System Usability Scale (SUS) | about 1 week after the end of the intervention
  Scores on the System Usability Scale (SUS) range from 0-100, with higher scores indicating greater usability (which is the desired outcome).
Acceptability as Assessed by the Acceptability E-Scale | about 1 week after the end of the intervention
  Scores on the Acceptability E-scale range from 6-30, with higher scores indicating greater acceptability (which is the desired outcome).
Feasibility as Assessed by Participation Rate | from the start of the intervention to the end of the intervention (6 weeks)
  Scores on the LaTrobe Social Communication Questionnaire (LCQ) range from 30-120, with lower score indicating less social communication impairment (which is the desired outcome).
Feasibility as Assessed by Attrition Rate | from the start of the intervention to the end of the intervention (6 weeks)

SECONDARY OUTCOMES:
Change in Social Communication as Assessed by the LaTrobe Communication Questionnaire (LCQ) | baseline, about 1 week after the end of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Hilary N Touchett, PhD(c), Principal Investigator — The University of Texas Health Science Center, Houston
Locations (2):
- United States (2):
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - TIRR Memorial Hermann, Houston, Texas

IPD SHARING:
Plan to Share IPD: No